CLINICAL TRIAL: NCT07043062
Title: Laparoscopic Versus Open Surgical Repair of Genitovesical Fistula in Females :ِ A Prospective Comparative Non Randomized Study
Brief Title: Laparoscopic Versus Open Surgical Repair of Genitovesical Fistula in Females
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Hassan Elshazly Khodary, Resident at Urology Department, Faculty of Medicine, South Valley University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Female Genitovesical fistula
Record Dates: First submitted 2025-05-21; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-08

CONDITIONS: Genitovesical Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of Laparoscopic Repair (Active Comparator): About 25 female patients suffering from Vesicovaginal fistula or Vesicouterine fistula and will be subjected to Laparoscopic repair of the fistula
  Interventions: Procedure: Open surgical Interference
- Group of Open Surgical Repair (Active Comparator): About 25 female patients suffering from Vesicovaginal fistula or Vesicouterine fistula and will be subjected to surgical repair of the fistula.
  Interventions: Procedure: Open surgical Interference

INTERVENTIONS:
Procedure: Open surgical Interference — to compare the outcomes of Laparoscopic repair versus Open surgical repair of Genitovesical fistula in females.
  Other Names: Laparoscopic Repair

SUMMARY:
Fistula is an abnormal passway that connects two organs or vessels that do not connect normally.

Genitourinary fistula refers to a fistula that occurs between reproductive tract organs (vagina, cervix, and uterus), and lower urinary tract (bladder, urethra, and pelvic ureters).

It is a serious condition which can significantly influence the biological and psychological condition of women, with a negative impact on the quality of life.

DETAILED DESCRIPTION:
Fistula is an abnormal passway that connects two organs or vessels that do not connect normally.

Genitourinary fistula refers to a fistula that occurs between reproductive tract organs (vagina, cervix, and uterus), and lower urinary tract (bladder, urethra, and pelvic ureters).

It is a serious condition which can significantly influence the biological and psychological condition of women, with a negative impact on the quality of life.

In developed countries, iatrogenic injury during hysterectomy or pelvic surgery is the primary cause of fistulae . However, the etiology differs in developing countries, being secondary to prolonged, obstructed, complicated labor.

Genitovesical fistulae are one of the most devastating complications in the urogynecology setting. The commonest type of these fistulae is the vesicovaginal fistula (VVF);the patients Suffering from continuous urinary leakage through the vagina and urinary smell, patients with VVF face hygienic, social, infectious, psychological, and sexual problems.

Vesicouterine fistulae (VUF) are not as common as VVF. In 1908, the first case was reported by Knipe , and later in 1957, Youssef reported on the classic symptoms of VUF. These symptoms included amenorrhea and cyclic hematuria, or menouria; known afterward as Youssef's syndrome. The prevalence of these fistulae is estimated to be 1-4% of all genitourinary fistulae.

Several options for the management of such fistulae have been discussed; these include conservative treatment with prolonged catheterization , open surgery, cysto-fulguration, endourology, and laparoscopy/robotic surgery. The decision-making is guided by the patient characteristics, etiology, and the experience of the treating surgeon.

Laparoscopy is of great advantage when compared to open surgery, including safe, effective, minimally invasive procedure, less postoperative pain, smaller incisions, lower blood loss, a shorter hospital stay, and faster recovery. It is associated with a lower incidence of postoperative complications, including infections and improper wound healing

ELIGIBILITY:
Inclusion Criteria:

* Females with Vesicovaginal fistula or Vesicouterine fistula.
* Timing of repair after 2-6 months of beginning of symptoms and signs of fistula.

Exclusion Criteria:

* Malignant , Recurrant or Post Radiation Genitovesical fistula.
* Females with congenital disease in Bladder ,Uterus or Vagina.
* Females with Vaginal or Uterine prolapse.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Treatment of Genitourinary fistula | From base line to 2 Months from the starting of the operation
  To examine the female patients whom suffering fromGenitourinary fistula, either by surgical interference or Laparoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aboalyosr Mohamed, Professor, Study Chair — Urology Department, Faculty of Medicine, South Valley University, Qena, Egypt
Locations (1):
- South Valley University Hospital, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided